CLINICAL TRIAL: NCT03156985
Title: Multi-center, Single Arm, Observational Study to Evaluate the Safety of Dapagliflozin in Type 2 Diabetes Mellitus Patients in China
Acronym: DONATE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1690R00027
Record Dates: First submitted 2017-05-16; First posted 2017-05-17 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
DONATE study is a multi-center, prospective cohort, single arm, observational study to be performed in 3000 Chinese type 2 diabetes mellitus (T2DM) patients recruited from 100 tier 2 or 3 hospitals, China.It is a drug intense monitoring study required by China Food and Drug Administration (CFDA) to assess the newly approved drug in at least 3000 patients within the first five years after commercial launch. The primary objective is to demonstrate the safety of dapagliflozin by assessment of the incidence of adverse events and serious adverse events during 6-month follow up in Chinese patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Provision of subject informed consent prior to any study specific procedures.
* Chinese, Female or male.
* T2DM diagnosed by physicians according to 2013 Chinese Guideline for Diabetes, ie. 1) Patients with typical syndrome and with a FPG ≥ 7.0mmol/L and/or random plasma glucose ≥ 11.1mmol/L; and/or, 2) patients without typical syndrome and with repeated FPG ≥ 7.0mmol/L and/or 2 hour post challenged plasma glucose ≥ 11.1mmol/L.
* Subjects who already took at least one dose of dapagliflozin, which is prescribed by physicians based on their clinical practice. The prescription of dapagliflozin is separated from the decision to be included in the current study or not.

Exclusion Criteria:

* Being unable to comply with study-specified procedures.
* Participating in any other clinical trial currently or during the last 3 months.
* Previous enrolment in the present study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: T2DM diagnosed by physicians according to 2013 Chinese Guideline for Diabetes and had been initiated the therapy of dapagliflozin by a physician (any licensed physician is qualified) and had taken at least one dose of dapagliflozin.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | within 6-months
  The adverse event will be collected and coded using latest version of MedDra. The incidence of adverse events will be presented using the number and percentages by System Organ Class and Preferred Term.

OTHER OUTCOMES:
Absolute change in HbA1c | 6 months
  Absolute change in HbA1c after the treatment with dapagliflozin
The proportion of patients achieving HbA1c less than 7.0% | 6 months
  The proportion of patients achieving HbA1c less than 7.0% after treatment with dapagliflozin that will be presented by percentage.
The absolute change in fasting plasma glucose (FPG) | 6 months
  The absolute change in FPG after treatment with dapagliflozin
The absolute change in postprandial plasma glucose (PPG) | 6 months
  The absolute change in PPG after treatment with dapagliflozin
The absolute change in body weight | 6 months
  The absolute change in body weight after treatment with dapagliflozin.
The absolute change in waist circumference | 6 months
  The absolute change in waist circumference after treatment with dapagliflozin.
The absolute change in blood pressure | 6 months
  The absolute change in blood pressure after treatment with dapagliflozin.
The incidence of interested adverse events | within 6 months
  The incidence of interested adverse events, including volume depletion, abnormal of blood electrolytes, polyuria, renal impairment, diabetic ketoacidosis, hepatic impairment, and hematuria, will be presented by number and percentage.

CONTACTS AND LOCATIONS:
Locations (51):
- China (51):
  - Research Site, Hefei, Anhui
  - Research Site, Huainan, Anhui
  - Research Site, Maanshan, Anhui
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Chongqing, Chongqing Municipality
  - Research Site, Lanzhou, Gansu
  - Research Site, Dongguan, Guangdong
  - Research Site, Foshan, Guangdong
  - Research Site, Guangzhou, Guangdong
  - Research Site, Huizhou, Guangdong
  - Research Site, Shenzhen, Guangdong
  - Research Site, Yingcheng, Guangdong
  - Research Site, Zhanjiang, Guangdong
  - Research Site, Zhaoqing, Guangdong
  - Research Site, Zhuhai, Guangdong
  - Research Site, Guilin, Guangxi
  - Research Site, Guiyang, Guizhou
  - Research Site, Shijiazhuang, Hebi
  - Research Site, Xingxiang, Henan
  - Research Site, Zhengzhou, Henan
  - Research Site, Wuhan, Hubei
  - Research Site, Changsha, Hunan
  - Research Site, Guankou, Hunan
  - Research Site, Hohhot, Inner Mongolia
  - Research Site, Kunshan, Jiangsu
  - Research Site, Lianyungang, Jiangsu
  - Research Site, Nanjing, Jiangsu
  - Research Site, Nantong, Jiangsu
  - Research Site, Qidong, Jiangsu
  - Research Site, Xuzhou, Jiangsu
  - Research Site, Yancheng, Jiangsu
  - Research Site, Dalian, Liaoning
  - Research Site, Shengyang, Liaoning
  - Research Site, Xining, Qinghai
  - Research Site, Xi'an, Shaanxi
  - Research Site, Jinan, Shandong
  - Research Site, Laizhou, Shandong
  - Research Site, Qingdao, Shandong
  - Research Site, Weifang, Shandong
  - Research Site, Zibo, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Taiyuan, Shanxi
  - Research Site, Nanchong, Sichuan
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Ürümqi, Xinjiang
  - Research Site, Kunming, Yunnan
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Ningbo, Zhejiang
  - Research Site, Ruian, Zhejiang
  - Research Site, Wenling, Zhejiang
  - Research Site, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Guo L, Wang J, Li L, Yuan L, Chen S, Wang H, Li T, Qi L, Yang H. A multicentre, prospective, non-interventional study evaluating the safety of dapagliflozin in patients with type 2 diabetes in routine clinical practice in China (DONATE). BMC Med. 2023 Jun 14;21(1):212. doi: 10.1186/s12916-023-02906-7. PMID 37316847
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1690R00027&attachmentIdentifier=ff77d148-dd44-46f0-8655-cff09ebd2010&fileName=DONATE_STUDY_REPORT_SYNOPSIS_EN_Update.pdf&versionIdentifier=